CLINICAL TRIAL: NCT04203784
Title: Meropenem and Piperacillin Plasma Concentrations During CRRT
Acronym: ABC2
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Petersson, Senior ICU Consultant, Karolinska University Hospital
Other Study IDs: K 2019-9604
Record Dates: First submitted 2019-11-03; First posted 2019-12-18 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Sepsis; Infection; Antibiotic; Renal Replacement Therapy; Hemolysis
MeSH Terms: conditions — Sepsis; Infections; Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Meropenem treated patients
  Interventions: Other: Plasma concentration measurements
- Piperacillin treated patients
  Interventions: Other: Plasma concentration measurements

INTERVENTIONS:
Other: Plasma concentration measurements — Plasma concentration measurements

SUMMARY:
This observational study reports meropenem and piperacillin plasma concentrations in patients treated with either antibiotic and simultaneous continuous renal replacement therapy (CRRT).

ELIGIBILITY:
Inclusion Criteria:

* patients treated in the study ICU and
* simultaneous CRRT and antibiotic treatment with either meropenem or piperacillin-tazobactam.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma antibiotic concentrations at mid and end of dosing interval | 1 week
  We vill report the measured plasma antibiotic concentrations at the mid and end of the dosing interval.
Plasma antibiotic concentrations at mid and end of dosing interval | 1 week
  The percentage of patients having a concentration above the highest MIC (minimal inhibitory concentration) breakpoint for pathogens considered susceptible for the antibiotic.
Relationships between plasma antibiotic concentrations and CRRT dose. | 1 week
  We will report the correlation between measured plasma concentrations of either antibiotic and the intensity of the CRRT treatment.
Influence of residual diuresis on the measured plasma antibiotic concentrations. | 1 week
  We will report the correlation between measured plasma concentrations of either antibiotic and residual diuresis.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided